CLINICAL TRIAL: NCT00402025
Title: Targeted Delivery of OncoVEX^GM-CSF by Endoscopic Ultrasound (EUS)-Guided Fine Needle Injection (FNI) in Patients With Irresectable Pancreatic Cancer: A Pilot Multinational Experiment on Safety and Proof of Concept
Brief Title: Talimogene Laherparepvec in Patients With Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioVex Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 005/04
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Results first posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Pancreatic Cancer
Keywords: Metastatic; Pancreas; Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis; Adenocarcinoma | interventions — talimogene laherparepvec

ARMS (1):
- Talimogene Laherparepvec (Experimental): Participants received 3 doses of talimogene laherparepvec administered by direct injection 3 weeks apart. At the discretion of the investigator, treatment with talimogene laherparepvec could continue beyond the third dose until week 15 in a regimen of at least 3 weeks between doses.
  Interventions: Biological: Talimogene Laherparepvec

INTERVENTIONS:
Biological: Talimogene Laherparepvec — Talimogene laherparepvec administered by direct injection into pancreatic tumors using EUS-guided FNI, up to a maximum of 4 mL per treatment.
  Other Names: OncoVEX^GM-CSF; T-VEC; IMLYGIC

SUMMARY:
The purpose of the study is to assess the safety of injections of talimogene laherparepvec into patients with pancreatic cancer that cannot be removed by surgery. The study will also test whether the injections are effective in treating the tumor.

DETAILED DESCRIPTION:
Talimogene laherparepvec is a conditionally replication competent herpes simplex type-1 virus designed for use in solid tumors. It has been specifically modified to replicate in tumors and to provide a local source of the immune-stimulating cytokine, granulocyte macrophage colony stimulating factor (GM-CSF). It is injected directly into cancer tumors and is believed to destroy tumor cells by direct infection of the tumor cells and an enhanced immune response due to the release of tumor antigens and GM-CSF expression.

This was an open-label, dose-escalation study evaluating the safety and efficacy of talimogene laherparepvec administered by direct injection into pancreatic tumors using endoscopic ultrasound (EUS)-guided fine needle injection (FNI). Only 1 tumor mass within the body and tail of the pancreas was injected in any participant. The protocol called for evaluation of 4 dosing regimens in sequential cohorts of participants; however, cohort 4 was not opened for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* cytological or histological proof of adenocarcinoma of the pancreas
* unresectable, locally advanced disease (isolated liver metastases are permitted)
* tumors of at least 1 cm diameter at screening
* measurable disease using Response Evaluation Criteria In Solid Tumors (RECIST) criteria
* failure of either standard therapy, OR any one of the following:

  * no alternative therapeutic of higher curative potential is available;
  * investigator determination that patient could not tolerate alternative therapeutic due to unacceptable toxicity; or,
  * patient refusal to be treated with available alternative therapeutic
* age > 18 years
* life expectancy > 3 months
* adequate bone marrow function as indicated by:

  * White blood cells (WBC) ≥ 3.0 x 10^9/L
  * platelets ≥ 100 x 10^9/L
  * hemoglobin ≥ 8.5 gm/dL
* adequate liver function as indicated by:

  * bilirubin < 1.5 x upper limit of normal (ULN)
  * alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 5 x ULN in case of presence of liver metastasis
  * ALT or AST < 2.5 x ULN in case of absence of liver metastasis
* adequate renal function as indicated by a serum creatinine level < 1.5 x ULN.
* adequate hemostasis indicated by international normalized ratio (INR) ≤ 1.5
* mentally, physically and geographically able to undergo treatment and follow-up
* provided written informed consent
* first patient in each cohort only: seropositive for herpes simplex virus type 1 (HSV1)

Exclusion Criteria:

* history of other malignancy within two years prior to screening, except for prostate cancer (T1c, T2ab with definitive treatment, prostate-specific antigen (PSA) < 1 ng/ml, and without ongoing hormone suppression) or adequately treated in situ carcinoma of the cervix, basal cell carcinoma, or squamous cell carcinoma of the skin
* cystic form of pancreatic cancer; microcystic disease may be eligible upon discussion with Medical Monitor
* Common Terminology Criteria for Adverse Events (CTCAE) version 3 grade 2 or greater clinical pancreatitis within 8 weeks prior to dosing with OncoVEX^GM-CSF
* other than metastases limited to the liver, imaging evidence of metastatic disease to any other organ or tissue
* any serious concomitant systemic disorder that would compromise the safety of the patient, at the discretion of the investigator
* evidence of compromised immune function including but not limited to:

  * clinically significant absolute lymphocyte count < Lower Limit of Normal (LLN)
  * known human immunodeficiency virus (HIV), acute or chronic active hepatitis B, or hepatitis C infection;
  * concurrently taking HIV antiviral medications (e.g. protease inhibitors, azidothymidine, etc.)
* received intravenous (IV), intramuscular (IM) or subcutaneous (SC) human gamma globulin within 6 months prior to dosing with OncoVEX^GM-CSF
* patients taking immunosuppressive agents (e.g. cyclosporine, tacrolimus, or oral or systemic corticosteroids at a dose of > 10 mg/day of prednisone or equivalent).
* pregnancy, lactation or lack of effective contraception in women of child-bearing potential (e.g., not post menopausal for > 2 years, or had tubal ligation); lack of effective contraception in men if the partner is of child-bearing potential; women must have been practicing an effective contraceptive method for at least three months prior to entry in to the trial (hormonal contraception or intrauterine device in conjunction with a barrier method); men must use a condom or be surgically sterilized
* patients with active bacterial or viral infections that require treatment with systemic antibiotics or antiviral agents within 2 weeks prior to the first dose of OncoVEX^GM-CSF); (note: patients with active cold sores or other HSV1 infections must wait until those lesions have crusted over before receiving OncoVEX^GM-CSF)
* surgery requiring general or spinal anesthesia within four weeks prior to dosing with OncoVEX^GM-CSF
* Treatment with an investigational agent within 4 weeks prior to the first dose of OncoVEX^GM-CSF
* serum carbohydrate antigen (CA)19.9 levels > 3000 U/mL at screening
* evidence of ascites on screening abdominal computed tomography (CT) scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil N Senzer, MD, Principal Investigator — Mary Crowley Medical Research Center; Robert Coffin, PhD, Study Director — BioVex Limited
Locations (3):
- United States (3):
  - UCI Medical Center, Orange, California
  - California Pacific Medical Center, San Francisco, California
  - Mary Crowely Medical Research Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled sequentially into each dose cohort.
Groups:
- Talimogene Laherparepvec 10⁴/ 10⁵ PFU/mL: Participants received 3 doses of talimogene laherparepvec; an initial dose of 10⁴plaque-forming units (PFU)/mL followed by 2 doses of 10⁵ PFU/mL, each 3 weeks apart.
  At the discretion of the investigator, treatment with talimogene laherparepvec could continue beyond the third dose until Week 15 in a regimen of at least 3 weeks between doses.
- Talimogene Laherparepvec 10⁵ / 10⁶ PFU/mL: Participants received 3 doses of talimogene laherparepvec; an initial dose of 10⁵ PFU/mL followed by 2 doses of 10⁶ PFU/mL, each 3 weeks apart.
  At the discretion of the investigator, treatment with talimogene laherparepvec could continue beyond the third dose until Week 15 in a regimen of at least 3 weeks between doses.
- Talimogene Laherparepvec 10⁶ / 10⁷ PFU/mL: Participants received 3 doses of talimogene laherparepvec; an initial dose of 10⁶ PFU/mL followed by 2 doses of 10⁷ PFU/mL, each 3 weeks apart.
  At the discretion of the investigator, treatment with talimogene laherparepvec could continue beyond the third dose until Week 15 in a regimen of at least 3 weeks between doses.
Period: Overall Study
Arm/Group | Talimogene Laherparepvec 10⁴/ 10⁵ PFU/mL | Talimogene Laherparepvec 10⁵ / 10⁶ PFU/mL | Talimogene Laherparepvec 10⁶ / 10⁷ PFU/mL
Started | 3 | 4 | 10
Completed | 1 | 1 | 0
Not Completed | 2 | 3 | 10
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Death | 0 | 1 | 5
Not completed — Disease Progression | 1 | 1 | 2
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Participant Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intention-to-Treat (ITT) population included all participants who received at least 1 dose of talimogene laherparepvec.
Groups:
- Talimogene Laherparepvec 10⁴/ 10⁵ PFU/mL: Participants received 3 doses of talimogene laherparepvec; an initial dose of 10⁴PFU/mL followed by 2 doses of 10⁵ PFU/mL, each 3 weeks apart.
  At the discretion of the investigator, treatment with talimogene laherparepvec could continue beyond the third dose until Week 15 in a regimen of at least 3 weeks between doses.
- Total: Total of all reporting groups
Arm/Group | Talimogene Laherparepvec 10⁴/ 10⁵ PFU/mL | Talimogene Laherparepvec 10⁵ / 10⁶ PFU/mL | Talimogene Laherparepvec 10⁶ / 10⁷ PFU/mL | Total
Number analyzed (Participants) | 3 | 4 | 10 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (10.97) | 63.8 (10.21) | 50.8 (6.68) | 54.5 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3 | 6
  Male | 3 | 1 | 7 | 11
Race/Ethnicity, Customized [Number; unit: participants]
  White | 2 | 3 | 8 | 13
  Black | 1 | 1 | 0 | 2
  Other | 0 | 0 | 2 | 2
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Scale used to assess how a patient's disease is progressing, how the disease affects the daily living abilities of the patient: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory, able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self care, confined to a bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  participants
    0 (Fully active) | 1 | 0 | 2 | 3
    1 (Restrictive but ambulatory) | 1 | 3 | 7 | 11
    2 (Ambulatory but unable to work) | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: A serious adverse event is defined as any untoward medical occurrence that at any dose results in death, is life threatening, requires hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, is an important and significant medical event that, based upon appropriate medical judgment, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed above.
Time Frame: From first dose of talimogene laherparepvec until 30 days after the last dose; the median duration of treatment was 44.0 days, 22.0 days, and 11.5 days in each group respectively.
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Talimogene Laherparepvec 10⁴/ 10⁵ PFU/mL | Talimogene Laherparepvec 10⁵ / 10⁶ PFU/mL | Talimogene Laherparepvec 10⁶ / 10⁷ PFU/mL
Number analyzed (Participants) | 3 | 4 | 10
participants
  Any adverse event | 3 | 4 | 10
  Serious adverse events | 2 | 3 | 9
  Deaths | 1 | 1 | 6
  Discontinued study treatment due to adverse event | 0 | 0 | 2

2. Secondary Outcome: Change From Baseline in Sum of Longest Diameters of Injected Tumors
Description: Spiral computed tomography (CT) scans were performed to assess tumors at screening and at Weeks 6, 12 and 18 after the initial dose.
Time Frame: Baseline and Week 6, 12 and 18
Population: ITT population with available data at each time point (indicated by "N").
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Talimogene Laherparepvec 10⁴/ 10⁵ PFU/mL | Talimogene Laherparepvec 10⁵ / 10⁶ PFU/mL | Talimogene Laherparepvec 10⁶ / 10⁷ PFU/mL
Number analyzed (Participants) | 3 | 4 | 10
mm
  Week 6 (N=2, 1, 4) | 2.5 (3.54) | 18.0 (NA) — Could not be calculated due to a sample size = 1 | -3.3 (12.42)
  Week 12 (N=1, 1, 0) | 0.0 (NA) — Could not be calculated due to a sample size = 1 | 18.0 (NA) — Could not be calculated due to a sample size = 1 | NA (NA) — Could not be calculated due to a sample size = 0
  Week 18 (N=2, 2, 1) | 11.5 (9.19) | 25.5 (10.61) | 37.0 (NA) — Could not be calculated due to a sample size = 1

3. Secondary Outcome: Number of Participants With Overall Objective Response
Description: Tumor response was assessed via CT scan by the investigator using Response Evaluation Criteria In Solid Tumors (RECIST) v1.0 guidelines. Objective response is defined as a complete response (CR) or partial response (PR).
  CR: Disappearance of all target and non-target lesions, normalization of tumor marker level and no new lesions and with confirmation no less than 4 weeks after the criteria for CR is first met.
  PR: At least a 30% decrease in the sum of longest diameters of target lesions taking as reference the baseline sum of the longest diameters, absence of non-target lesion progression, and no new lesions. These criteria must be confirmed no less than 4 weeks after they are first met.
Time Frame: Every 6 weeks until 12 weeks after the last dose; the median duration of treatment was 44.0 days, 22.0 days, and 11.5 days in each group respectively.
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Talimogene Laherparepvec 10⁴/ 10⁵ PFU/mL | Talimogene Laherparepvec 10⁵ / 10⁶ PFU/mL | Talimogene Laherparepvec 10⁶ / 10⁷ PFU/mL
Number analyzed (Participants) | 3 | 4 | 10
participants | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Talimogene Laherparepvec Detected in Blood and Urine
Description: Samples of blood and urine collected before and up to 24 hours after dosing were tested for the presence of talimogene laherparepvec deoxyribonucleic acid (DNA) using a validated quantitative polymerase chain reaction (qPCR) assay.
Time Frame: Treatment Day 1 predose and 2, 6, 12 and 24 hours postdose, and Week 3 and 6 at (predose and 2 hours postdose.
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Talimogene Laherparepvec 10⁴/ 10⁵ PFU/mL | Talimogene Laherparepvec 10⁵ / 10⁶ PFU/mL | Talimogene Laherparepvec 10⁶ / 10⁷ PFU/mL
Number analyzed (Participants) | 3 | 4 | 10
participants
  Blood | 0 | 4 | 1
  Urine | 1 | 2 | 4

5. Primary Outcome: Number of Participants Positive for Anti-herpes Simplex Virus-1 (HSV-1) Antibodies
Description: Anti-HSV-1 antibodies were detected using an enzyme-linked immunosorbent assay (ELISA).
Time Frame: Week 0 (Day 1, predose) and Week 3
Population: ITT population with available antibody results (indicated by N)
Measure: Number; unit: participants
Arm/Group | Talimogene Laherparepvec 10⁴/ 10⁵ PFU/mL | Talimogene Laherparepvec 10⁵ / 10⁶ PFU/mL | Talimogene Laherparepvec 10⁶ / 10⁷ PFU/mL
Number analyzed (Participants) | 3 | 4 | 10
participants
  Baseline (predose) (N= 3, 3, 8) | 2 | 3 | 6
  Week 3 (N=3, 3, 6) | 3 | 3 | 6

6. Secondary Outcome: Change From Baseline in Pain Intensity
Description: Pain was assessed by the participant using a validated Visual Analog Scale (VAS) pain assessment instrument. A single 10-cm line was used with the leftmost end (0 cm) representing "no pain" and the rightmost end (10 cm) representing "worst pain". The distance was measured from the leftmost part of the scale to the mark made by the participant indicating pain level.
Time Frame: Baseline and Weeks 3 and 6
Population: ITT population with available VAS data; this assessment was added in the third protocol amendment and change from baseline could only be assessed for participants in cohort 3.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Talimogene Laherparepvec 10⁴/ 10⁵ PFU/mL | Talimogene Laherparepvec 10⁵ / 10⁶ PFU/mL | Talimogene Laherparepvec 10⁶ / 10⁷ PFU/mL
Number analyzed (Participants) | 0 | 0 | 6
cm
  Week 3 (N=0, 0, 6) |  |  | 1.250 (2.456)
  Week 6 (N=0, 0, 4) |  |  | 2.575 (3.305)

ADVERSE EVENTS:
Time Frame: From first dose until study discontinuation; the median (minimum, maximum) duration of time in the study was 13.0 (6.0, 32.1) weeks, 5.5 (0.1, 21.0) weeks and 3.1 (0.1,16.1) weeks in each treatment group respectively.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Talimogene Laherparepvec 10⁴/ 10⁵ PFU/mL | Talimogene Laherparepvec 10⁵ / 10⁶ PFU/mL | Talimogene Laherparepvec 10⁶ / 10⁷ PFU/mL
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/4 | 9/10
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talimogene Laherparepvec 10⁴/ 10⁵ PFU/mL (N=3) | Talimogene Laherparepvec 10⁵ / 10⁶ PFU/mL (N=4) | Talimogene Laherparepvec 10⁶ / 10⁷ PFU/mL (N=10)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 1
BRADYCARDIA (Cardiac disorders) | 0 | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 0 | 0 | 1
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 2
ASCITES (Gastrointestinal disorders) | 1 | 0 | 3
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1
CHEST PAIN (General disorders) | 0 | 0 | 1
DISEASE PROGRESSION (General disorders) | 0 | 1 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 0 | 3
BACTERAEMIA (Infections and infestations) | 1 | 0 | 0
ACIDOSIS (Metabolism and nutrition disorders) | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 1
METASTATIC PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 1 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
HYPOTENSION (Vascular disorders) | 0 | 0 | 1
SUPERIOR MESENTERIC ARTERY SYNDROME (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Talimogene Laherparepvec 10⁴/ 10⁵ PFU/mL (N=3) | Talimogene Laherparepvec 10⁵ / 10⁶ PFU/mL (N=4) | Talimogene Laherparepvec 10⁶ / 10⁷ PFU/mL (N=10)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 2 | 3
SPLENOMEGALY (Blood and lymphatic system disorders) | 0 | 0 | 1
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 1 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1
HYPOTHYROIDISM (Endocrine disorders) | 0 | 0 | 1
DRY EYE (Eye disorders) | 0 | 0 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 0 | 3
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 6
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0 | 0
ANORECTAL DISORDER (Gastrointestinal disorders) | 0 | 0 | 1
ASCITES (Gastrointestinal disorders) | 1 | 0 | 5
COLITIS (Gastrointestinal disorders) | 0 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 1 | 5
DIARRHOEA (Gastrointestinal disorders) | 2 | 0 | 2
FLATULENCE (Gastrointestinal disorders) | 1 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1
GASTROINTESTINAL OEDEMA (Gastrointestinal disorders) | 0 | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 1 | 1
HIATUS HERNIA (Gastrointestinal disorders) | 0 | 0 | 1
ILEUS (Gastrointestinal disorders) | 0 | 0 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 2 | 0 | 4
PANCREATITIS (Gastrointestinal disorders) | 0 | 0 | 1
STEATORRHOEA (Gastrointestinal disorders) | 1 | 0 | 0
STOMACH DISCOMFORT (Gastrointestinal disorders) | 1 | 0 | 0
VOMITING (Gastrointestinal disorders) | 1 | 1 | 3
ASTHENIA (General disorders) | 0 | 0 | 1
CATHETER RELATED COMPLICATION (General disorders) | 0 | 0 | 1
CHEST PAIN (General disorders) | 0 | 0 | 1
CHILLS (General disorders) | 0 | 0 | 1
FATIGUE (General disorders) | 0 | 0 | 1
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 1 | 1
OEDEMA PERIPHERAL (General disorders) | 1 | 0 | 0
PAIN (General disorders) | 1 | 0 | 2
PYREXIA (General disorders) | 0 | 1 | 3
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 0 | 1 | 0
BILE DUCT STENOSIS (Hepatobiliary disorders) | 1 | 0 | 0
JAUNDICE (Hepatobiliary disorders) | 1 | 1 | 0
SEASONAL ALLERGY (Immune system disorders) | 1 | 0 | 0
ABDOMINAL INFECTION (Infections and infestations) | 0 | 1 | 0
CANDIDIASIS (Infections and infestations) | 0 | 1 | 0
INFECTION (Infections and infestations) | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
AMMONIA INCREASED (Investigations) | 0 | 1 | 0
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 | 0 | 1
BLOOD AMYLASE INCREASED (Investigations) | 1 | 0 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 1 | 0
BLOOD CREATINE INCREASED (Investigations) | 1 | 0 | 0
LIPASE INCREASED (Investigations) | 1 | 0 | 0
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 1 | 0
WEIGHT DECREASED (Investigations) | 0 | 0 | 1
ANOREXIA (Metabolism and nutrition disorders) | 0 | 0 | 2
CACHEXIA (Metabolism and nutrition disorders) | 0 | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 2 | 0 | 4
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 1 | 0 | 1
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 0 | 1
MEMORY IMPAIRMENT (Nervous system disorders) | 0 | 0 | 1
SOMNOLENCE (Nervous system disorders) | 0 | 1 | 0
SYNCOPE VASOVAGAL (Nervous system disorders) | 0 | 0 | 1
AGITATION (Psychiatric disorders) | 0 | 0 | 1
ANXIETY (Psychiatric disorders) | 0 | 0 | 1
DELIRIUM (Psychiatric disorders) | 0 | 0 | 1
DEPRESSION (Psychiatric disorders) | 0 | 0 | 1
HALLUCINATION (Psychiatric disorders) | 0 | 0 | 2
INSOMNIA (Psychiatric disorders) | 0 | 0 | 3
URINARY RETENTION (Renal and urinary disorders) | 0 | 1 | 0
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
HERNIA REPAIR (Surgical and medical procedures) | 0 | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 3
HYPOTENSION (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.